CLINICAL TRIAL: NCT00103038
Title: NCI-Sponsored Multi-Disciplinary Study for MR Imaging of Intravenous Superparamagnetic Crystalline Particle Ferumoxytol in Primary High-Grade Brain Tumors and/or Cerebral Metastases
Brief Title: Ferumoxytol in Improving MR Imaging in Patients With High-Grade Brain Tumors or Cerebral Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Edward Neuwelt, Professor, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00000813; NCI-2015-00226 (Other: National Cancer Institute); ONC-03095-LX (Other: OHSU Knight Cancer Institute); IRB00000813 (Other: OHSU Knight Cancer Institute); R01CA137488 (NIH); NCT00980720 (obsolete NCT alias)
Record Dates: First submitted 2005-02-07; First posted 2005-02-08 (Estimated); Results first posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-05

CONDITIONS: Central Nervous System Lymphoma; Malignant Glioma; Metastatic Malignant Neoplasm in the Brain
MeSH Terms: conditions — Glioma; Brain Neoplasms | interventions — Ferrosoferric Oxide; Gadolinium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (ferumoxytol, gadolinium, DCE-MRI, DSC-MRI) (Experimental): Study patients: adult patients with high grade primary malignant brain tumors or with known or suspected brain metastases from histologically confirmed primary cancer
  Study procedures: patients will receive IV ferumoxytol (maximum dose 4 mg/kg, over at least 15 minutes) beginning approximately 15 seconds after start of 3T DSC-MRI and GBCA IV approximately 1 minute and 50 seconds after start of 3T DCE-MRI on day 1. Patients will also undergo MRI without contrast at baseline (before and on day 2. Imaging with ferumoxytol, GBCA and without contrast repeats every 3 weeks for a total of 6 more imaging sessions over up to 5 years.
  3 Tesla Magnetic Resonance Imaging: Undergo 3T MRI
  Dynamic Contrast-Enhanced Magnetic Resonance Imaging: Undergo 3T DCE-MRI
  Dynamic Susceptibility Contrast-Enhanced Magnetic Resonance Imaging: Undergo 3T DSC-MRI
  Ferumoxytol: Given IV
  Gadolinium: Given IV
  MRI-Based Angiogram: Undergo MRA
  Interventions: Procedure: 3 Tesla Magnetic Resonance Imaging; Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging; Procedure: Dynamic Susceptibility Contrast-Enhanced Magnetic Resonance Imaging; Drug: Ferumoxytol; Drug: Gadolinium; Procedure: MRI-Based Angiogram

INTERVENTIONS:
Procedure: 3 Tesla Magnetic Resonance Imaging — Undergo 3T MRI
  Other Names: 3 Tesla MRI; 3T MRI
Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging — Undergo 3T DCE-MRI
  Other Names: DCE MRI; DCE-MRI; DYNAMIC CONTRAST ENHANCED MRI
Procedure: Dynamic Susceptibility Contrast-Enhanced Magnetic Resonance Imaging — Undergo 3T DSC-MRI
  Other Names: Dynamic Susceptibility Contrast-Enhanced MRI
Drug: Ferumoxytol — Given IV
  Other Names: Feraheme; FERUMOXYTOL NON-STOICHIOMETRIC MAGNETITE
Drug: Gadolinium — Given IV
  Other Names: Gd
Procedure: MRI-Based Angiogram — Undergo MRA
  Other Names: Magnetic Resonance Angiogram; MRA

SUMMARY:
This clinical trial studies magnetic resonance imaging (MRI) using a contrast imaging agent ferumoxytol (ferumoxytol non-stoichiometric magnetite) in improving viewing tumors in patients with high-grade brain tumors or cancer that has spread to the brain. Diagnostic procedures, such as MRI, may help find and diagnose brain tumors and find out how far the disease has spread. The contrast imaging agent ferumoxytol non-stoichiometric magnetite consists of small iron particles taken by the blood stream to the brain and to the area of the tumor. It may help visualize the blood flow going through the tumor better than the standard substance gadolinium-based contrast agent.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Investigate the utility of ferumoxytol and gadolinium-based contrast agent (GBCA) for improved imaging biomarkers of malignant brain tumors in a single imaging session by comparing dynamic susceptibility contrast (DSC) determined relative cerebral blood volume (rCBV) and dynamic contrast enhancement (DCE) determined vascular permeability (derived transfer coefficient [Ktrans]).

SECONDARY OBJECTIVES:

I. Compare and evaluate magnetic resonance angiography (MRA) with ferumoxytol between different time points.

II. Assess number and size of tumors imaged. III. Assess tumor vascularity. IV. Assess histology and electron microscopy (EM) on tissue samples. V. Assess differences in subjects with prior therapy versus (vs.) no prior therapy (radiation and/or chemotherapy).

VI. Assess the long term imaging characteristics of different tumors using DSC and DCE.

OUTLINE:

Patients receive ferumoxytol non-stoichiometric magnetite intravenously (IV) beginning approximately 15 seconds after start of 3T DSC-MRI and GBCA IV approximately 1 minute and 50 seconds after start of 3T DCE-MRI on day 1. Patients also undergo MRI without contrast at baseline and on day 2. Imaging with ferumoxytol, GBCA, and without contrast repeats every 3 weeks for a total of 6 more imaging sessions over up to 5 years.

After completion of study, patients are followed up at approximately 4-6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have either radiological or established histological diagnosis of the following general categories:

  * High-grade glioma/central nervous system (CNS) lymphoma or
  * Brain metastases
* Previously untreated subjects must have a lesion on an imaging study
* Post treatment subjects will have radiographic abnormalities that may or may not be recurrent tumor
* Subjects agree to be contacted 4-6 weeks after each study visit
* Subjects, or their legal guardian, must sign a written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization in accordance with institutional guidelines
* Sexually active women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) prior to study treatment and for the duration of study treatment; should a female become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Pre-imaging radiological scans/studies must be performed approximately 16 weeks prior to study entry; but not less than 24 hours prior

Exclusion Criteria:

* Subjects with clinically significant signs of uncal herniation, such as acute pupillary enlargement, rapidly developing motor changes (over hours), or rapidly decreasing level of consciousness, are not eligible
* Subjects with known allergic or hypersensitivity reactions to parenteral iron, parenteral dextran, parenteral iron-dextran, or parenteral iron-polysaccharide preparations (Ferumoxytol Investigator's Drug Brochure, 2012); subjects with significant drug or other allergies or autoimmune diseases may be enrolled at the investigator's discretion
* Subjects who are pregnant or lactating or who suspect they might be pregnant
* Subjects who require monitored anesthesia for MRI scanning
* Subjects with renal insufficiency; glomerular filtration rate (GFR) < 50
* Subjects who have a contraindication for MRI: metal in their bodies (a cardiac pacemaker or other incompatible device), are severely agitated, or have an allergy to gadolinium (Gd) contrast material
* Subjects with known hepatic insufficiency or cirrhosis
* Human immunodeficiency virus (HIV)-positive subjects on combination antiretroviral therapy are ineligible
* Subjects with known or suspected iron overload (genetic hemochromatosis or history of multiple transfusions)
* Subjects with three or more drug allergies from separate drug classes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2004-06-04 (Actual); Primary Completion 2016-05-10 (Actual); Study Completion 2016-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Neuwelt, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Malignant Brain Tumor Patients Undergoing Brain MRI (With Both Ferumoxytol and Gadolinium): Study patients: adult patients with high grade primary malignant brain tumors or with known or suspected brain metastases from histologically confirmed primary cancer
  Study procedures: patients will receive IV ferumoxytol (maximum dose 4 mg/kg, over at least 15 minutes) beginning approximately 15 seconds after start of 3T DSC-MRI and GBCA IV approximately 1 minute and 50 seconds after start of 3T DCE-MRI on day 1. Patients will also undergo MRI without contrast at baseline (before and on day 2. Imaging with ferumoxytol, GBCA and without contrast repeats every 3 weeks for a total of 6 more imaging sessions over up to 5 years.
  3 Tesla Magnetic Resonance Imaging: Undergo 3T MRI
  Dynamic Contrast-Enhanced Magnetic Resonance Imaging: Undergo 3T DCE-MRI
  Dynamic Susceptibility Contrast-Enhanced Magnetic Resonance Imaging: Undergo 3T DSC-MRI
  Ferumoxytol: Given IV
  Gadolinium: Given IV
  MRI-Based Angiogram: Undergo MRA
Period: Overall Study
Arm/Group | Malignant Brain Tumor Patients Undergoing Brain MRI (With Both Ferumoxytol and Gadolinium)
Started | 155
Completed | 142
Not Completed | 13
Not completed — Withdrawal by Subject | 8
Not completed — Screen failure | 3
Not completed — Death | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Malignant Brain Tumor Patients Undergoing Brain MRI (With Both Ferumoxytol and Gadolinium)
Number analyzed (Participants) | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.71 (13.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 150
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 147
  More than one race | 0
  Unknown or Not Reported | 2
Type of brain malignancy [Count of Participants; unit: Participants]
  Glioblastoma | 67
  Anaplastic Astrocytoma | 19
  Anaplastic Oligodendroglioma | 19
  Primary CNS Lymphoma | 4
  Brain metastasis | 18
  Other | 17
  Unknown | 11

OUTCOME MEASURES:

1. Primary Outcome: Utility of Femumoxytol and Gadolinium Based Contrast Agents for Improved Imaging Biomarkers of Malignant Brain Tumors in a Single Session by Comparing Dynamic Contrast Enhanced Determined Vascular Permeability (Ktrans)
Description: Appropriate descriptive statistics (mean, standard deviation, minimum, median, and maximum) will be estimated for the imaging parameters Ktrans. Frequency distributions of each parameter will also be described to assess normality. Pearson's correlation coefficients will be estimated to describe potential relationships among these various measures.
Time Frame: Assessed after each visit for up to 6 imaging sessions (up to 5 years)
Population: Software to derive K trans values from acquired images is not available and enhancement comparison between gadolinium and ferumoxytol K trans values is not possible to date.
Arm/Group | Malignant Brain Tumor Patients Undergoing Brain MRI (With Both Ferumoxytol and Gadolinium)
Number analyzed (Participants) | 0

2. Primary Outcome: Utility of Ferumoxytol and Gadolinium Based Contrast Agents for Improved Imaging Biomarkers of Malignant Brain Tumors in a Single Imaging Session by Comparing Dynamic Susceptibility Contrast (DSC) Determined Relative Cerebral Blood Volume (rCBV) Maps.
Description: Compare rCBV measurements in regions of interest obtained from ferumoxytol DSC-MRI with gadolinium based contrast agent (GBCA) MR images to evaluate vascular properties of brain tumors. CBV maps were generated by applying tracer kinetic model to the first pass of the contrast bolus. Voxelwise CBV maps were coregistered to T1 weighted images and then normalized by dividing by the mean of normal appearing white matter CBV in the same region in the contralateral hemisphere. RCBV values (as the area under the signal intensity curve, normalized by the area under the curve for the control region) were obtained. Values range from 0 (low intensity) to 180 (highest intensity).
Time Frame: Summarized after completion of up to 6 imaging sessions (up to 5 years)
Measure: Mean (Full Range); unit: Values on a scale
Groups:
- Malignant Brain Tumor Patients Undergoing Brain MRI: Study patients: adult patients with high grade primary malignant brain tumors or with known or suspected brain metastases from histologically confirmed primary cancer
  Study procedures: patients will receive IV ferumoxytol (maximum dose 4 mg/kg, over at least 15 minutes) beginning approximately 15 seconds after start of 3T DSC-MRI and GBCA IV approximately 1 minute and 50 seconds after start of 3T DCE-MRI on day 1. Patients will also undergo MRI without contrast at baseline (before and on day 2. Imaging with ferumoxytol, GBCA and without contrast repeats every 3 weeks for a total of 6 more imaging sessions over up to 5 years.
  3 Tesla Magnetic Resonance Imaging: Undergo 3T MRI
  Dynamic Contrast-Enhanced Magnetic Resonance Imaging: Undergo 3T DCE-MRI
  Dynamic Susceptibility Contrast-Enhanced Magnetic Resonance Imaging: Undergo 3T DSC-MRI
  Ferumoxytol: Given IV
  Gadolinium: Given IV
  MRI-Based Angiogram: Undergo MRA
Arm/Group | Malignant Brain Tumor Patients Undergoing Brain MRI
Number analyzed (Participants) | 12
Values on a scale
  Peritumor area gadolinium rCBV | 146 [0 to 180]
  Peritumor area ferumoxytol rCBV | 136 [0 to 180]
  Tumor area gadolinium rCBV | 39 [0 to 180]
  Tumor area ferumoxytol rCBV | 54 [0 to 180]

3. Secondary Outcome: Compare Number and Size of Tumors Imaged With Ferumoxytol and Gadolinium Based Contrast Agents (Cube Root Volume)
Description: We analyzed 193 sets of post-gadoteriol and 24 hours post-ferumoxytol T1 weighted scans from 58 patient with high grade glioma. Enhancement volumes normalized to normal appearing white matter were calculated with histogram analysis. Enhancement cube root volumes were compared between the two contrast agents. Ferumoxytol and gadolinium enhanced MR images were obtained from each participant.
Time Frame: Summarized after completion of up to 6 imaging sessions (up to 5 years)
Population: 58 participants had both appropriate ferumoxytol and gadolinium scans available for analysis for this outcome.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: MR images/scans
Groups:
- Malignant Brain Tumor Patients Undergoing Brain MRI- Gadolinium-enhanced MRI; Malignant Brain Tumor Patients Undergoing Brain- Ferumoxytol-enhanced MRI: Study patients: adult patients with high grade primary malignant brain tumors or with known or suspected brain metastases from histologically confirmed primary cancer
  Study procedures: patients will receive IV ferumoxytol (maximum dose 4 mg/kg, over at least 15 minutes) beginning approximately 15 seconds after start of 3T DSC-MRI and GBCA IV approximately 1 minute and 50 seconds after start of 3T DCE-MRI on day 1. Patients will also undergo MRI without contrast at baseline (before and on day 2. Imaging with ferumoxytol, GBCA and without contrast repeats every 3 weeks for a total of 6 more imaging sessions over up to 5 years.
  3 Tesla Magnetic Resonance Imaging: Undergo 3T MRI
  Dynamic Contrast-Enhanced Magnetic Resonance Imaging: Undergo 3T DCE-MRI
  Dynamic Susceptibility Contrast-Enhanced Magnetic Resonance Imaging: Undergo 3T DSC-MRI
  Ferumoxytol: Given IV
  Gadolinium: Given IV
  MRI-Based Angiogram: Undergo MRA
Arm/Group | Malignant Brain Tumor Patients Undergoing Brain MRI- Gadolinium-enhanced MRI | Malignant Brain Tumor Patients Undergoing Brain- Ferumoxytol-enhanced MRI
Number analyzed (Participants) | 58 | 58
Number analyzed (MR images/scans) | 193 | 193
mm | 21.71 (6.396) | 18.71 (6.884)

4. Secondary Outcome: Compare Number and Size of Tumors Imaged With Ferumoxytol and Gadolinium Based Contrast Agents (Signal Intensity)
Description: We analyzed 193 sets of post-gadoteriol and 24 hours post-ferumoxytol T1 weighted scans from 58 patient with high grade glioma. Signal intensities normalized to normal appearing white matter were calculated with histogram analysis. Signal intensities were compared between the two contrast agents. Ferumoxytol and gadolinium enhanced MR images were obtained from each participant. Signal intensities were normalized to the signal intensity value of non-enhancing voxels inside the manual ROI (the relative complement of the final mask in Q, i.e. Q \ [A ∩ B ∩ C]). Higher values in signal intensity indicated increased image enhancement.
Time Frame: Summarized after completion of up to 6 imaging sessions (up to 5 years)
Population: 58 participants had both appropriate ferumoxytol and gadolinium scans available for analysis for this outcome.
Measure: Mean (Standard Deviation); unit: ratio
Units Other Than Participants: Images
Arm/Group | Malignant Brain Tumor Patients Undergoing Brain MRI- Gadolinium-enhanced MRI | Malignant Brain Tumor Patients Undergoing Brain- Ferumoxytol-enhanced MRI
Number analyzed (Participants) | 58 | 58
Number analyzed (Images) | 193 | 193
ratio | 1.36 (0.107) | 1.26 (0.108)

5. Secondary Outcome: Overall Survival in Participants With Pseudoprogression With or Real Tumor Progression Using Ferumoxytol Enchanced Perfusion MRI
Description: We evaluated overall survival in patients with pseudopregression or real tumor progression by using relative cerebral blood volume values on ferumoxytol enhanced perfusion MRIs.
Time Frame: Assessed after each visit for up to 6 imaging sessions (up to 5 years)
Population: 68 participants had appropriate ferumoxytol scans available for analysis for this outcome.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Malignant Brain Tumor Patients Undergoing Brain MRI
Number analyzed (Participants) | 68
months
  Median survival in patients with pseudoprogression seen on Fe-MRI: number analyzed (Participants) | 24
  Median survival in patients with pseudoprogression seen on Fe-MRI | 34.7 [20.3 to 54.1]
  Median survival in patients with real progression seen on Fe-MRI: number analyzed (Participants) | 44
  Median survival in patients with real progression seen on Fe-MRI | 13.4 [11.1 to 19.5]

ADVERSE EVENTS:
Time Frame: Subjects were evaluated for adverse events approximately 4-6 weeks after each study visit, up to 5 years.
Description: Patients are monitored for adverse events in the scanning unit for the entire MRI time and 30 minutes after the final infusion of ferumoxytol An additional phone follow up visit was performed 4-6 weeks after each imaging session to focus on any new adverse events
Groups:
- Malignant Brain Tumor Patients Undergoing Brain MRI (With Both Ferumoxytol and Gadolinium): Study patients: adult patients with high grade primary malignant brain tumors
  Study procedures: patients will receive IV ferumoxytol (maximum dose 4 mg/kg, over at least 15 minutes) beginning approximately 15 seconds after start of 3T DSC-MRI and GBCA IV approximately 1 minute and 50 seconds after start of 3T DCE-MRI on day 1. Patients will also undergo MRI without contrast at baseline (before and on day 2. Imaging with ferumoxytol, GBCA and without contrast repeats every 3 weeks for a total of 6 more imaging sessions over up to 5 years.
  3 Tesla Magnetic Resonance Imaging: Undergo 3T MRI
  Dynamic Contrast-Enhanced Magnetic Resonance Imaging: Undergo 3T DCE-MRI
  Dynamic Susceptibility Contrast-Enhanced Magnetic Resonance Imaging: Undergo 3T DSC-MRI
  Ferumoxytol: Given IV
  Gadolinium: Given IV
  MRI-Based Angiogram: Undergo MRA
Arm/Group | Malignant Brain Tumor Patients Undergoing Brain MRI (With Both Ferumoxytol and Gadolinium)
All-Cause Mortality (participants affected / at risk) | 119/155
Serious Adverse Events (participants affected / at risk) | 0/152
Other Adverse Events (participants affected / at risk) | 12/152
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Malignant Brain Tumor Patients Undergoing Brain MRI (With Both Ferumoxytol and Gadolinium) (N=152)
Hypertension (Cardiac disorders) | 12 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes